CLINICAL TRIAL: NCT01815996
Title: Identify Clinical Conditions That Increase Circulating DNA Levels
Acronym: BARDA II
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 407-2012; IRB201702171 (Other: University of Florida)
Record Dates: First submitted 2013-03-12; First posted 2013-03-21 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Pulmonary Embolism; Myocardial Infarction; Autoimmune Disease
Keywords: Pregnancy; pulmonary embolism; myocardial infarction; autoimmune disease; healthy controls
MeSH Terms: conditions — Pulmonary Embolism; Myocardial Infarction; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4-5 ml of blood will be processed and the plasma will be divided into 150 μl aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pregnant Women: Females between the age of 18-80 who are pregnant
  One time blood draw to look at patient's DNA
  Interventions: Other: One time blood draw to look at patient's DNA
- Pulmonary Embolism Patients: Male and Female patients that have suffered a pulmonary embolism within the past 48 hours
  One time blood draw to look at patient's DNA
  Interventions: Other: One time blood draw to look at patient's DNA
- Myocardial Patients: Male and Female patients who have myocardial infarction in the past 48 hours.
  One time blood draw to look at patient's DNA
  Interventions: Other: One time blood draw to look at patient's DNA
- Autoimmune Patients: Male and Female patients that have been diagnosed with an Autoimmune disease
  One time blood draw to look at patient's DNA
  Interventions: Other: One time blood draw to look at patient's DNA
- Healthy Controls: Self-declared healthy adults (men and women).
  One time blood draw to look at patient's DNA
  Interventions: Other: One time blood draw to look at patient's DNA

INTERVENTIONS:
Other: One time blood draw to look at patient's DNA — One time blood draw to look at patient's DNA

SUMMARY:
The investigators are developing a test that is expected to measure the amount of radiation a patient has been exposed to after a nuclear bomb. The investigator will do this by measuring the DNA in the patients blood from cells killed by the radiation.

Many diseases and medical conditions can put DNA in the blood. The investigator needs to know how much DNA in order to better interpret our radiation detection test. Therefore, the investigator is collecting blood from several patients with different diseases or medical conditions and also healthy volunteers to measure their DNA content.

Patients that will be included in this study are pregnant women, patients who have suffered a pulmonary embolism within the past 48 hours, patients who have suffered from myocardial infarction in the past 48 hours, patients with autoimmune diseases and health patients.

DETAILED DESCRIPTION:
The investigator will collect 8 mL (one and one half teaspoons) of blood one time only. The investigator may also collect the patient's past medical history, test results and disease treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be adults in one of the following categories:

   * Pregnant
   * Suffered a pulmonary embolism within the past 48 hours
   * Myocardial infarction in the past 48 hours
   * Diagnosed with an autoimmune disease
   * Adults age 18-80
   * Self-declared healthy adults
2. Patients must be willing to undergo a blood draw
3. Patients must provide study-specific informed consent prior to study entry

Exclusion Criteria:

1. Patients not meeting the above inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeking healthy volunteers, pregnant women, patients who recently suffered a heart attach or pulmonary embolism, and patiebts with autoimmune disease. Patients who are health individuals will also be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Different diseases will be analysed for the levels of DNA circulating in the blood | blood will be tested up to 1 year after collection
  To determine what medical conditions and disease states might increase circulating DNA levels at a magnitude similar to whole body irradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Okunieff, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Davis Cancer Center, Gainesville, Florida, United States